CLINICAL TRIAL: NCT04268264
Title: Effect of Incremental Introduction of Dialysis Versus Standard Care in Patients With End-stage Renal Disease: a Feasibility Study
Brief Title: A Feasibility Study to Test the Acceptability, Tolerance and Safety of Incremental Haemodialysis
Acronym: ENDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2338
Record Dates: First submitted 2019-11-14; First posted 2020-02-13 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Renal Failure; Hemodialysis Complication; Morality
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Will receive trial intervention, Incremental haemodialysis (n=20)
  Interventions: Procedure: Incremental haemodialysis
- Control arm (Other): Historical controls. Matched controls from database of historical patients receiving conventional, three times weekly haemodialysis treatment (n=40)
  Interventions: Procedure: Conventional haemodialysis

INTERVENTIONS:
Procedure: Incremental haemodialysis — twice weekly haemodilysis at the start, gradually building up to full dose dialysis over a period of 15 weeks
  Arms: Treatment arm
Procedure: Conventional haemodialysis — three times weekly 4-hour long haemodialysis sessions from the start
  Arms: Control arm

SUMMARY:
This feasibility study tests if patients find incremental HD acceptable, whether they tolerate the treatment as planned and to evaluate its safety. Over a period of 18-months, 20 participants will be recruited in to the study who are about to start HD therapy for ESRD. The participants will start HD incrementally (incremental HD group) reaching full dose HD over a period of approximately 15 weeks. The outcomes will be compared to a cohort of 40 matched patients who previously started HD in the conventional manner (historical controls, conventional HD group).

All patients will be followed-up for 6 months after first dialysis. Participants will be reviewed regularly during this time, and will undergo laboratory and bed-site monitoring tests. Acceptability and tolerance will be tested by documenting the numbers and percentages of patients who agree to participate and continue in the study. Patients who decline the invitation to join the study will be given the opportunity to express their reasons for declining to go on incremental HD (they will not play further part in the study). The safety of incremental HD will be tested by comparing the rates of pre-defined safety events in the incremental HD vs. conventional HD groups.

The impact of incremental HD on patients' residual renal function will be monitored using serial 24-hour urine collections, bio-impedance testing will be conducted to estimate changes in fluid load, measurements of quality-of-life will be undertaken by using patient KDQOL-SF v1.3 questionnaires. These tests will be repeated at regular intervals. Blood tests for estimation of residual renal function and markers of renal anemia, bone disease and cardiac load will be performed at regular intervals and will be compared between the two groups (incremental HD vs. conventional HD groups). These measurements will help in the evaluation of impact of incremental HD on patients' health and well-being. The completion rates of these tests will provide important information about whether they should be included in a future larger trial of incremental HD. Participants undergoing incremental HD will be invited to take part in semi-structured interviews aimed at exploring patients' experiences of receiving incremental HD and their participation in the study.

Data from this study will be used to test if it is feasible to use deaths (or a combination of deaths and cardiovascular events) as the main outcome measure in a future definitive trial on incremental HD. The data should enable a sample-size calculation for a future full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* patients with CKD-5 who are about to start planned HD
* At least 3 months of prior specialist renal follow-up at the time of starting HD
* Able to meet all the study requirements
* Written signed informed consent.

Exclusion Criteria:

* Age < 18
* No prior contact with nephrologists for > 3 months
* Cross-over in to HD from peritoneal dialysis
* Currently undergoing HD therapy
* Any condition which in the opinion of the investigator makes the participant unsuitable for entry in to the study
* Participation in an interventional study in the preceding 6 weeks
* History of myocardial infarction in the preceding 3 months
* Inability to provide informed consent
* Inability to comply with the study schedule and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability: Recruitment rate | 6 months
  What proportion of eligible patients were recruited in to the trial?
Tolerance: Retention rate | 6 months
  What proportion of participants completed treatment as planned
Completion rates of non-routine tests | 6 months
  Completion rates of the non-routine tests a) the 24-hour urine collections, b) six-minute walk test, c) bio-impedance testing and d) quality of life questionnaires

SECONDARY OUTCOMES:
Mortality and cardiovascular event rates | 6 months
  Differences in mortality, and the composite of mortality and major cardiovascular events, between the interventional and control groups.
Mechanistic 1: Rate of loss of residual renal function in the interventional group | 6 months
  Differences in renal urea clearance (in millilitres/min) from baseline
Mechanistic 2:Changes in fluid load | 6 months
  Differences in overhydration volume (as measured through bio-impedance testing)
Mechanistic 3:Quality of life | 6 months
  Changes in quality of life scores (using KDQOL-SF v 1.3) from baseline
Mechanistic 4: Anaemia control | 6 months
  Changes in haemoglobin levels from baseline
Mechanistic 5: Parathyroid hormone control | 6 months
  Changes in serum Parathyroid hormone, calcium and phosphate levels from baseline
Mechanistic 6: Cardiac load | 6 months
  Changes in serum NT-proBNP measurements from baseline
Safety 1: pre dialysis hyperkalaemia | 6 months
  Number of events: pre-dialysis hyperkalaemia (6.5 mmol/l or above)
Safety 2: severe hypertension | 6 months
  Number of events: severe pre-dialysis hypertension (systolic BP > 180 and/or diastolic BP > 110 mmHg)
Safety 3: Inter-dialytic weight gain | 6 months
  Number of events: interdialytic weight gain of greater than 4 kg

CONTACTS AND LOCATIONS:
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided